CLINICAL TRIAL: NCT06839807
Title: Adequately Diagnosing Total Knee Arthroplasty Loosening: A Randomized Controlled Trial Evaluating the AtMoves Knee System in a Routine Clinical Setting
Brief Title: DIGITAL-KNEE Study: Adequately Diagnosing Total Knee Arthroplasty Loosening by Evaluating the AtMoves Knee System in a Routine Clinical Setting
Acronym: DigitalKnee
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Sint Maartenskliniek (Other)
Responsible Party: Principal Investigator, Leendert Blankevoort, Associate professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DIGITAL-KNEE - 2024.0590
Record Dates: First submitted 2025-01-07; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Aseptic Loosening; Aseptic Loosening of Prosthetic Joint; Aseptic Loosening of Orthopaedic Hardware; Knee Arthroplasty, Total; Total Knee Arthroplasty (Replacement)
Keywords: Aseptic loosening of total knee prosthesis; Aseptic loosening; Total knee arthroplasty; Aseptic loosening of prosthetic joint; Knee arthroplasty

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (RCT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention: AtMoves Knee System group (Experimental): The intervention group will undergo a CT-scan using the AtMoves Knee System. They are allowed to undergo the diagnostic pathway determined by their treating orthopedic surgeon.
  Interventions: Device: AtMoves Knee System
- Control: usual care/diagnostics (No Intervention): The control group is not allowed to undergo a CT-scan using the AtMoves Knee System. They will undergo the diagnostic pathway determined by their treating orthopedic surgeon.

INTERVENTIONS:
Device: AtMoves Knee System — The AtMoves Knee Stystem is a loading device that is able to exert force in varus and valgus. when these forces are applied during a CT-scan micromotions of the tibial component of the total knee prosthesis can be detected.
  Arms: Intervention: AtMoves Knee System group

SUMMARY:
The goal of the clinical trial is to evaluate the efficacy of the AtMoves Knee System in the clinical diagnostic process of aseptic loosening in patients with a knee prosthesis. The main question it aims to answer is:

Does the use of the AtMoves Knee System reduce the percentage of failed outcomes? A "failed outcome" is defined as a change in the patient-reported Knee injury and Osteoarthritis Outcome Score (KOOS-PS) that is lower than the minimal clinically important difference at 12 months.

Researchers will compare two groups: The first group will undergo an additional CT scan using the AtMoves Knee System. The second group will not undergo these scans. Both groups are allowed to undergo additional diagnostic measures. Researchers will compare the percentage of "failed outcomes" between these groups.

During the one-year follow-up, participants in both groups will be asked to fill out questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Subjects must have underwent either unilateral or bilateral TKA surgery.
* Aseptic loosening is one of the differential diagnoses of the treating orthopaedic surgeon
* The treating Orthopaedic Surgeon is uncertain of the diagnosis after anamnesis, physical examination and conventional x-ray.
* The surgeon wants additional examinations or additional imaging to arrive at the diagnosis and proposal for treatment.
* Subjects must be capable of giving informed consent and must be willing to undergo examination with the AtMoves Knee System.

Exclusion Criteria:

* A clear other cause for complaints other than aseptic loosening (e.g. septic loosening, neuropathic pain, non-consolidated peri-prosthetic fracture of the bone around the TKA)
* Surgical interventions of the index knee in the year prior to the start of the complaints associated with TKA loosening.
* Posttraumatic or congenital deformation of the leg for which the loading device does not fit.
* Pregnancy or suspected pregnancy.
* Unable or unwilling to understand or sign the informed consent for this study and to undergo examination with the AtMoves Knee System.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Failed Outcome | 12 months
  The primary outcome measure is the status of the outcome of the treatment as "failed outcome" at 12 months as determined by a change in KOOS-PS (Knee Injury and Osteoarthritis Outcome Score-Physical function Short form) that is less than the minimal clinically important difference (MCID) compared to baseline KOOS-PS (MCID is set to 15). The KOOS-PS gives a score from 0-100 with higher scores reflecting better physical function.

SECONDARY OUTCOMES:
Revision surgery | 12 months
  The number of participants between the two arms that undergo revision surgery in the 12 months follow up period despite the initial decision (based on the diagnostic pathway) to not perform revision surgery.
Number of Diagnostic activities | until the final diagnostic decision (up to six months)
  The number and types of diagnostic activities until the final diagnostic treatment decision is made in all subjects
Cost of diagnostic activities | Upon the final diagnostic decision (up to six months).
  The cost of diagnostic activities until the final diagnostic treatment decision is made in all subjects. For cost-effectiveness evaluation. This will be measured using a version of the iMTA Medical Consumption Questionnaire (iMCQ).
Medical consumption after diagnosis | 1 Year
  Medical consumption costs after final diagnosis and treatment until the end of follow-up (1 year). Measured using the iMTA Medical Consumption Questionnaire at 1 year follow-up.
Societal productivity loss after diagnosis | 1 Year
  Societal productivity loss after final diagnosis and treatment until the end of follow-up (1 year). Measured using the iMTA Productivity Cost Questionnaire at 1 year follow-up.
Subject satisfaction intervention group | Day of CT-scan using the AtMoves Knee system (day 0)
  Satisfaction of undergoing the AtMoves Knee System, measured in trial subjects randomized in the intervention arm. Measured by a short questionnaire including pain during- and after the scan (10 point numeric rating scale), subjective satisfaction of the scan (10 point numeric rating scale), and open field option for any comments on satisfaction on the day of the scan.

CONTACTS AND LOCATIONS:
Locations (7):
- Netherlands (7):
  - St. Maartenskliniek, Nijmegen, Gelderland
  - Zuyderland Ziekenhuis, Heerlen, Limburg
  - Amphia ziekenhuis, Breda, North Brabant
  - Amsterdam UMC, Amsterdam, North Holland
  - OCON, Hengelo, Overijsel
  - NoordWest Ziekenhuisgroep, Alkmaar
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg

IPD SHARING:
Plan to Share IPD: No
IPD will not be made pubicly available but can be obtained upon request at the study's sponsor. When a valid reason for the re-use of study data is provided, a Data Sharing Agreement can be set up.

REFERENCES:
- [Background] Buijs GS, Kievit AJ, Ter Wee MA, Magg C, Dobbe JGG, Streekstra GJ, Schafroth MU, Blankevoort L. Non-invasive quantitative assessment of induced component displacement can safely and accurately diagnose tibial component loosening in patients: A prospective diagnostic study. Knee Surg Sports Traumatol Arthrosc. 2025 Jan;33(1):274-285. doi: 10.1002/ksa.12299. Epub 2024 May 31. PMID 38819937